CLINICAL TRIAL: NCT03070353
Title: Dextran, a Plasma Expander, Offers New Hope for Patients With Decompensated Liver Cirrhosis and Acute Kidney Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Abhasnee Sobhonslidsuk, Associate professor, Ramathibodi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID 11-57-21
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Cirrhosis, Liver; AKI
Keywords: Cirrhosis; AKI; Albumin; Dextran
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — Dextrans

STUDY DESIGN:
Intervention Model Description: Focus on clinical response after receiving treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dextran 40 (Experimental): Dextran 40 infusion
  Interventions: Drug: Dextran 40

INTERVENTIONS:
Drug: Dextran 40 — Dextran-40 infusion with the dose of 1 g/kg/day (10 ml/kg/day) for 2 days.
  Other Names: Colloidal plasma expander

SUMMARY:
A pilot study of Dextran-40 infusion in patients with decompensated cirrhosis presenting with AKI

DETAILED DESCRIPTION:
A pilot study of Dextran-40 infusion in decompensated cirrhotic patients complicating with AKI. Dextran-40® was administered at 1 g/kg/day for two days. AKI reversal was defined when serum creatinine was < 1.5 mg/dL. Albumin infusion was given if AKI reversal did not occur.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated cirrhosis with acute kidney injury
* Ager over 18 years old

Exclusion Criteria:

* Having chronic kidney disease, severe heart or lung disease, severe sepsis
* Pregnant
* Receiving nephrotoxic agents
* Having history of allergic to Dextran

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
AKI reversal | 2 weeks
  Reducing creatinine to below 1.5 mg/dl

SECONDARY OUTCOMES:
Mortality | 1 year
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Abhasnee Sobhonslidsuk, MD, Principal Investigator — Ramathibodi Hospital

IPD SHARING:
Plan to Share IPD: No
IPD will be provided if directly contact with investigator

REFERENCES:
- [Result] Niemi TT, Miyashita R, Yamakage M. Colloid solutions: a clinical update. J Anesth. 2010 Dec;24(6):913-25. doi: 10.1007/s00540-010-1034-y. Epub 2010 Oct 17. PMID 20953964